CLINICAL TRIAL: NCT06068439
Title: A Phase III Multi-center Randomized Placebo-controlled Study of the Protective Effect of Low-dose Aspirin on Renal Function in Patients With Early Diabetic
Brief Title: Study of the Protective Effect of Low-dose Aspirin on Renal Function in Patients With Early Diabetic Nephropathy
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SZNK2
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Nephropathy Type 2
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated group (Experimental)
  Interventions: Drug: Acetylsalicylic Acid
- Comparator group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic Acid — aspirin 50 mg/d to be taken after dinner (in nonfasting conditions)
  Arms: Treated group
Drug: Placebo — Placebo 50 mg/d to be taken after dinner (in nonfasting conditions)
  Arms: Comparator group

SUMMARY:
This is a multicenter, randomized, placebo-controlled study to evaluate the effectiveness and safety of low-dose aspirin (50 mg/day) in renal and cardiac function protection in people with diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* 1.Voluntarily sign informed consent;2.Meet the diagnosis of diabetic nephropathy: In the case of identifying diabetes as the cause of kidney damage and excluding chronic kidney disease caused by other causes, at least one of the following is present:①. In the case of excluding interference factors, at least 2 UACR≥30mg/g or UAER≥30mg/24h (≥20ug/min) in 3 tests within 3~6 months. ②. eGFR<60ml/min/(1.73m2)-1 for more than 3 months. ③. Renal biopsy consistent with pathological changes of DKD;3.DKD staging is 3 and before，eGFR>30ml/min/(1.73m2)-1；

Exclusion Criteria:

* (1) History of cardiovascular or cerebrovascular events (defined by the patient's medical history and/or instrumental examination results); (2)Insufficient glycemic control (i.e., glycated hemoglobin ≥8%); (3) Uncontrolled blood pressure despite taking antihypertensive drugs (≥140/≥85mmHg); (4) Previous major bleeding (i.e., intracranial hemorrhage); (5) Previous gastrointestinal ulcers; (6) Clinical diagnosis of type 1 diabetes mellitus (diagnosis of diabetes mellitus and use of insulin before age 35);(7) Patients with CKDG4 or G5 (i.e., eGFR<30 mL/min/1.73 m2 or dialysis) ;(8) chronic active infection or; (9) evidence of malignancy within the past 5 years. Patients with tumour disease in situ who are successfully treated only by local resection can be included in the study (including non-melanoma skin cancer in situ); (10) Autoimmune diseases; (11) Persistent arrhythmias requiring anticoagulation therapy (i.e., atrial fibrillation). In this category, isolated ventricular/supraventricular presystoles; (12) Use of NSAIDs or other antiplatelet drugs in the past 30 days; (13) cirrhosis of any etiology; (14) use of anticoagulants; (15) Life expectancy less than 1 year; (16) Known aspirin allergy; (17) Known pregnancy; and (18) Severe mental illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
decline of renal function | 3YEARS
  The aim of the study is to evaluate the decline of renal function, as assessed by absolute change in eGFR, calculated as the difference between eGFR at 3 years and baseline eGFR, in T2DM patients receiving low-dose aspirin (50 mg/d) or lacebo.

SECONDARY OUTCOMES:
The rapid decline in renal function | 3YEARS
  The rapid decline in renal function, defined as a reduction of eGFR ≥5 mL/min at 1 year
Change of renal function class | 3YEARS
  Change of renal function class (from G1 to G2, from G2 to G3a, and so on) at 3 years, dialysis, or transplantation